CLINICAL TRIAL: NCT04587934
Title: Time to Accurate Heart Rate on Neonatal Outcomes
Acronym: GE-EKG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: GE Healthcare (Industry); Sharp Mary Birch Hospital for Women & Newborns (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GE-EKG
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Premature Infant; Extremely Low Birth Weight; Extreme Prematurity
Keywords: electrocardiogram; Neonatal Resuscitation; resuscitation of premature infants
MeSH Terms: conditions — Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iRes Warmer with ResusView (Experimental): iRes Warmer with ResusView program with experimental electrocardiogram monitor will be used for heart rate monitoring in the first 10 minutes of life during routine care and and/or neonatal resuscitation.
  Interventions: Device: iRes Warmer with ResusView
- iRes Warmer without ResusView (Active Comparator): An external non-experimental electrocardiogram monitor will be used for heart rate monitoring in the first 10 minutes of life during routine care and and/or neonatal resuscitation.
  Interventions: Other: iRes Warmer without ResusView

INTERVENTIONS:
Device: iRes Warmer with ResusView — Rapid heart rate display utilizing optimized ECG algorithm in iRes Warmer in babies delivered between 23+0 and 32+6 weeks estimated gestational age
  Other Names: Panda Bed with ECG Feature
  Arms: iRes Warmer with ResusView
Other: iRes Warmer without ResusView — Electrocardiogram monitoring using external ECG monitor in babies delivered between 23+0 and 32+6 weeks estimated gestational age
  Other Names: Standard of Care
  Arms: iRes Warmer without ResusView

SUMMARY:
The goal of this trial is to compare the time to first heart rate displayed for iRes Warmer with ResusView and using iRes Warmer without ResusView when used in the resuscitation (e.g. Cardiopulmonary resuscitation or breathing assistance) of premature newborns (23 to 32+6 weeks gestation).

DETAILED DESCRIPTION:
This is a prospective interventional randomized control trial. Infants born between 23+0 and 32+6 estimated gestational age will be randomized using a computer generate allocation sequence stratified by gestational age. Randomization cards will be placed in opaque envelopes. For the intervention group, the care team will use the Panda iRes Warmer with ResusView Bed during resuscitation interventions in the first 10 minutes of life. During use of the iRes-warmer, standard nursing care of an infant on a radiant warmer will be followed. Participants assigned to the control group will receive interventions using the same model Panda bed without ResusView. There is no minimum time for monitoring, and the maximum time depends on clinical determination for use of heart rate feature for each resuscitation event. Data including the infant's gestational age, Electrocardiogram lead type and activities that occurred during resuscitation will be recorded for the first 10 minutes of life.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are delivered to mothers over the age of 16 years of age
* Infants delivered at 23+0 to 32+6 weeks estimated gestational age based on the best obstetric estimate at the time of delivery.
* Infants without known congenital malformations prior to delivery
* Antenatal consent

Exclusion Criteria:

* Infants who are delivered to mothers under the age of 16 years of age
* Known congenital anomalies of newborn prior to delivery
* Cardiac defects other than small Ventricular septum defect and Patent ductus arteriosus
* Multiples
* Declined consent
* iRes Warmer with ResusView not available at time of delivery

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, particularly data that underlie the results reported in this article after deidentification will be available with other researchers, including data dictionaries for meta-analysis.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 36 months following article publication
Access Criteria: Data and publication are available at clinicaltrials.gov
URL: https://pubmed.ncbi.nlm.nih.gov/34715091/

REFERENCES:
- [Background] Katheria A, Arnell K, Brown M, Hassen K, Maldonado M, Rich W, Finer N. A pilot randomized controlled trial of EKG for neonatal resuscitation. PLoS One. 2017 Nov 3;12(11):e0187730. doi: 10.1371/journal.pone.0187730. eCollection 2017. PMID 29099872
- [Background] Johnson PA, Schmolzer GM. Heart Rate Assessment during Neonatal Resuscitation. Healthcare (Basel). 2020 Feb 23;8(1):43. doi: 10.3390/healthcare8010043. PMID 32102255
- [Background] Neonatal Resuscitation. Vol. 7th edition. 2016, Elk Grove Village, IL: American Academy of Pediatrics.
- [Derived] Katheria AC, Morales A, Shashank S, Rich WD, Finer NN. A Pilot Randomized Trial of Heart Rate Monitoring Using Conventional Versus a New Electrocardiogram Algorithm during Neonatal Resuscitation at Birth. J Pediatr. 2022 Mar;242:245-247.e1. doi: 10.1016/j.jpeds.2021.10.037. Epub 2021 Oct 27. PMID 34715091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women who are dated by their earliest ultrasound scan or last menstrual period at 230/7 to 326/7 weeks of gestational age were identified, recruited, and consented from the labor and delivery floor or perinatal special care unit at Sharp Mary Birch Hospital Women & Newborns from February 2021 through June 2021.
Period: Overall Study
Arm/Group | iRes Warmer With ResusView | iRes Warmer Without ResusView
Started | 19 | 23
Completed | 19 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: all consented and enrolled in study
Groups:
- Total: Total of all reporting groups
Arm/Group | iRes Warmer With ResusView | iRes Warmer Without ResusView | Total
Number analyzed (Participants) | 19 | 23 | 42
Age, Continuous [Mean (Standard Deviation); unit: weeks gestational age at birth] | 28 (3) | 28 (3) | 28 (3)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 9 | 8 | 17
    Male | 10 | 15 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 23 | 42

OUTCOME MEASURES:

1. Primary Outcome: Time to Heart Rate Display in iRes Warmer With Resusview
Description: Measure time from birth to heart rate displayed on monitor following lead placement
Time Frame: Birth to 10 minutes of life
Population: All with available electrocardiogram data and prenatal consent
Measure: Mean (Standard Deviation); unit: seconds from time of birth
Arm/Group | iRes Warmer With ResusView | iRes Warmer Without ResusView
Number analyzed (Participants) | 19 | 23
seconds from time of birth | 16 (11) | 50 (50)

2. Secondary Outcome: Time to First Change in Fraction of Inspired Oxygen
Description: Measure time from birth to first increase or decrease in fraction of inspired oxygen from ECG lead placement
Time Frame: Birth to 10 minutes of life
Population: all subject with available electrocardiogram and fraction of inspired oxygen with consent prior to birth
Measure: Mean (Standard Deviation); unit: seconds from time of birth
Arm/Group | iRes Warmer With ResusView | iRes Warmer Without ResusView
Number analyzed (Participants) | 19 | 23
seconds from time of birth | 160 (140) | 175 (79)

3. Secondary Outcome: Time to First Change in Airway Pressure
Description: Measure time from birth to first increase or decrease in airway pressure from ECG lead placement
Time Frame: Birth to 10 minutes of life
Measure: Mean (Standard Deviation); unit: seconds from time of birth
Arm/Group | iRes Warmer With ResusView | iRes Warmer Without ResusView
Number analyzed (Participants) | 19 | 23
seconds from time of birth | 215 (204) | 100 (69)

4. Secondary Outcome: Time to Initiation of Positive Pressure Ventilation (PPV)
Description: Measure time from birth to start of PPV following first heart rate display
Time Frame: Birth to 10 minutes of life
Population: all with available electrocardiogram data and resuscitation intervention details
Measure: Mean (Standard Deviation); unit: seconds from time of birth
Arm/Group | iRes Warmer With ResusView | iRes Warmer Without ResusView
Number analyzed (Participants) | 19 | 23
seconds from time of birth | 58 (22) | 139 (79)

5. Other Pre Specified Outcome: Time of Electrode Placement
Description: Measure time from birth to application of Electrocardiogram electrodes from time of birth
Time Frame: Birth to 10 minutes of life
Population: all with electrocardiogram lead placement during resuscitation
Measure: Mean (Standard Deviation); unit: seconds from time of birth
Arm/Group | iRes Warmer With ResusView | iRes Warmer Without ResusView
Number analyzed (Participants) | 19 | 23
seconds from time of birth | 96 (24) | 112 (36)

6. Other Pre Specified Outcome: EKG Waveform Displayed by Rapid EKG Algorithm During Resuscitation
Description: Identify if a cardiac rhythm is recognized by Electrocardiogram monitor algorithm and displays a waveform during resuscitation (Yes/No)
Time Frame: Birth to 10 minutes of life
Population: all with electrocardiogram lead placement
Measure: Count of Participants; unit: Participants
Arm/Group | iRes Warmer With ResusView | iRes Warmer Without ResusView
Number analyzed (Participants) | 19 | 23
Participants | 19 | 23

7. Other Pre Specified Outcome: Time to Rhythm Recognition
Description: Measure at what time the Warmer displays the baby's cardiac rhythm
Time Frame: Birth to 10 minutes of life
Population: all with electrocardiogram data
Measure: Mean (Standard Deviation); unit: seconds from time of EKG lead placement
Arm/Group | iRes Warmer With ResusView | iRes Warmer Without ResusView
Number analyzed (Participants) | 19 | 23
seconds from time of EKG lead placement | 111 (28) | 161 (56)

ADVERSE EVENTS:
Time Frame: birth to 10 minutes of life
Description: Research/clinical staff collected information about resuscitation interventions for each participant at the time of birth
Arm/Group | iRes Warmer With ResusView | iRes Warmer Without ResusView
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 0/19 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT04587934/Prot_000.pdf